CLINICAL TRIAL: NCT00998400
Title: Cognitive-behavioral Treatment of Depression in Patients With Acute Coronary Syndrome
Brief Title: Treatment of Depression in Acute Coronary Syndrome (ACS) Patients
Acronym: TREATED-ACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Collaborators: Compagnia di San Paolo (Other)
Responsible Party: Principal Investigator, Chiara Rafanelli, Professor, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008.1263
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Results first posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-01

CONDITIONS: Depression
Keywords: Cognitive-behavioral treatment; Well-being therapy; Depression; Demoralization; Acute coronary syndrome
MeSH Terms: conditions — Depression; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clinical Management (No Intervention): Control group
- CBT + WBT (Experimental): Patients treated with Cognitive-Behavioral Therapy in combination with Well-Being Therapy and lifestyle modification
  Interventions: Behavioral: CBT in combination with WBT and life style modification

INTERVENTIONS:
Behavioral: CBT in combination with WBT and life style modification — CBT involves several essential features: identifying and correcting inaccurate thoughts associated with depressed feelings (cognitive restructuring); helping patients to engage more often in enjoyable activities (behavioral activation); enhancing problem-solving skills; providing instruction and guidance in specific strategies for solving problems. The techniques included in WBT may be used in overcoming impairments in environmental mastery, purpose in life, personal growth, autonomy, self-acceptance and positive relations with others. CM will consist of reviewing the patients' clinical status, and providing the patient with support and advice if necessary.
  Other Names: Cognitive-behavioural therapies
  Arms: CBT + WBT

SUMMARY:
Emotional states of depression in association with ischemic heart diseases, such as myocardial infarction or unstable angina, are risk factors for subsequent cardiac events and mortality. However, the only psychological intervention trial attempting to reduce cardiac risk in depressed ACS patients showed that changes in depression did not translate into improved survival. Such intervention did not address issues such as lifestyle modification and improvement in psychological well-being, which were found to affect individual vulnerability to medical disease. Our research group has developed a well-being enhancing psychotherapeutic strategy, well-being therapy (WBT), which has been validated in a number of clinical trials. The aim of this project is to evaluate the efficacy of cognitive behavioral treatment (CBT) together with lifestyle modification and WBT in reducing cardiac risk in depressed and/or demoralized ACS patients compared to a standard clinical procedure of patients' management, the clinical management (CM). The same protocol will be carried out in two centres (Bologna and Torino). 100 patients after a first episode of myocardial infarction or unstable angina, meeting DSM-IV criteria for depressive disorders and DCPR criteria for demoralization will be randomized to one of two treatment groups: 1) CBT supplemented by lifestyle modification and WBT; 2) CM. In both groups, treatment will consist of twelve, 45-minute sessions once a week. A two-year follow-up will be performed. It is expected that psychological treatment may significantly decrease cardiac morbidity and mortality at follow-up compared to clinical management. The findings may entail considerable preventive implications and possible large reductions in health costs.

DETAILED DESCRIPTION:
The same protocol will be carried out in the two participating centres (Maggiore Hospital in Bologna and San Giovanni Battista Hospital in Torino).

Participants will be patients recovering from a first episode of acute myocardial infarction or unstable angina. Myocardial infarction will be documented by cardiac symptoms (presence of acute chest, epigastric, neck, jaw, or arm pain or discomfort or pressure without apparent non- cardiac source) and signs (acute congestive heart failure or cardiogenic shock in the absence of non-CHD causes) associated with ECG findings (characteristic evolutionary ST-T changes or new Q waves) and/or cardiac biomarkers (blood measures of myocardial necrosis, specifically CK, CK-MB, CK-MBm, or troponin, cTn). Instable angina will be documented by cardiac symptoms (chest pain lasting less than 20 minutes) with likely ECG findings (ST-segment depression and abnormal T-wave) in absence of myocardial necrosis biomarkers.

Medically eligible patients involved in the study have to meet, when screened 30 days after their index event, the inclusion criteria

ELIGIBILITY:
Inclusion Criteria:

* a current diagnosis of at least one of the following: major or minor depression, dysthymia according to DSM-IV criteria, and demoralization according to DCPR criteria
* Mini-Mental State Examination score higher than 24
* written informed consent provided by the patient to participate

Exclusion Criteria:

* history of bipolar disorder (DSM-IV criteria)
* major depression with psychotic features
* history of substance abuse or dependency during the previous 12 months
* serious suicide risk
* current use of antidepressants
* current treatment with any form of psychotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-09; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Rafanelli, MD, Ph.D, Principal Investigator — Department of Psychology, University of Bologna
Locations (2):
- Italy (2):
  - Maggiore Hospital, Bologna
  - Molinette Hospital, Torino

REFERENCES:
- [Derived] Tully PJ, Ang SY, Lee EJ, Bendig E, Bauereiss N, Bengel J, Baumeister H. Psychological and pharmacological interventions for depression in patients with coronary artery disease. Cochrane Database Syst Rev. 2021 Dec 15;12(12):CD008012. doi: 10.1002/14651858.CD008012.pub4. PMID 34910821

RESULTS

PARTICIPANT FLOW:
Groups:
- CBT/WBT: Patients treated with Cognitive-Behavioral Therapy in combination with Well-Being Therapy and lifestyle modification
  CBT in combination with WBT and life style modification: CBT involves several essential features: identifying and correcting inaccurate thoughts associated with depressed feelings (cognitive restructuring); helping patients to engage more often in enjoyable activities (behavioral activation); enhancing problem-solving skills; providing instruction and guidance in specific strategies for solving problems. The techniques included in WBT may be used in overcoming impairments in environmental mastery, purpose in life, personal growth, autonomy, self-acceptance and positive relations with others.
- Clinical Management: Clinical management - CM (control group)
  Clinical management entails the same amount of time and attention from a professional figure than the experimental group, but specific interventions were proscribed. Such form of active control consisted of empathic listening, reviewing patients' clinical status, distress and worries, and encouragement of treatment adherence.
Period: Overall Study
Arm/Group | CBT/WBT | Clinical Management
Started | 50 | 50
Completed | 48 | 48
Not Completed | 2 | 2
Not completed — Lack of interest/motivation | 1 | 2
Not completed — Logistical problems | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- CBT/WBT: Patients treated with Cognitive-Behavioral Therapy in combination with Well-Being Therapy and lifestyle modification (expertimental group)
  CBT involves several essential features: identifying and correcting inaccurate thoughts associated with depressed feelings (cognitive restructuring); helping patients to engage more often in enjoyable activities (behavioral activation); enhancing problem-solving skills; providing instruction and guidance in specific strategies for solving problems. The techniques included in WBT may be used in overcoming impairments in environmental mastery, purpose in life, personal growth, autonomy, self-acceptance and positive relations with others.
- Total: Total of all reporting groups
Arm/Group | CBT/WBT | Clinical Management | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.64 (9.99) | 60.02 (10.94) | 58.83 (10.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 12 | 31
  Male | 31 | 38 | 69
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 50 | 50 | 100
Marital Status [Count of Participants; unit: Participants]
  Single | 4 | 7 | 11
  Married | 33 | 36 | 69
  Separated | 5 | 4 | 9
  Divorced | 2 | 1 | 3
  Widow/Widower | 6 | 2 | 8
Occupation [Count of Participants; unit: Participants]
  Employed | 34 | 24 | 58
  Unemployed | 1 | 4 | 5
  Retired | 13 | 19 | 32
  Homemaker | 2 | 3 | 5
Education [Count of Participants; unit: Participants]
  Primary school | 5 | 5 | 10
  Middle school | 16 | 18 | 34
  High school | 19 | 25 | 44
  University | 8 | 1 | 9
  Post-graduate education | 2 | 1 | 3
Type of ACS [Count of Participants; unit: Participants]
  STEMI acute myocardial infarction | 33 | 33 | 66
  NSTEMI acute myocardial infarction | 14 | 13 | 27
  Unstable angina | 3 | 4 | 7
GRACE index [Mean (Standard Deviation); unit: percent probability] — The Global Registry of Acute Coronary Events (GRACE) risk index is calculated during hospital admission and provides an estimate of the probability of cardiac mortality both during hospitalization and within 6 months from hospital discharge in patients with acute coronary syndrome (ACS).
  In order to calculate the GRACE risk index, the following data are needed: age, heart rate, systolic blood pressure, creatinine level, Killip class, cardiac arrest at admission, ST-segment deviation and elevated enzymes/markers.
  percent probability
    Probability of Death In-hospital (%) | 3.51 (8.58) | 4.56 (7.90) | 4.03 (8.22)
    Probability of Death Post-discharge to 6 Months (% | 6.60 (11.60) | 8.69 (10.57) | 7.64 (11.09)
Symptom Questionnaire [Mean (Standard Deviation); unit: scores on a scale] — Kellner's Symptom Questionnaire (SQ) is a 92-item self-report questionnaire, which yields 4 main scales including 23 items each: "depression", "anxiety", "hostility-irritability" and "somatization". This instrument helps the identification of self-perceived subclinical psychological distress. Answers are dichotomous (YES/NO or TRUE/FALSE) and rated with 0 or 1, therefore each scale score may range from 0 to 23. The higher the total score, the higher the psychological distress.
  scores on a scale
    Anxiety | 8.60 (4.73) | 7.24 (4.67) | 7.92 (4.73)
    Depression | 7.92 (4.77) | 6.90 (4.87) | 7.41 (4.82)
    Somatization | 9.82 (5.65) | 7.82 (5.12) | 8.82 (5.46)
    Hostility | 4.70 (4) | 5.34 (4.36) | 5.02 (4.17)
Psychological Well-Being scales [Mean (Standard Deviation); unit: scores on a scale] — The Psychological Well-Being scales (PWB), an 84-item questionnaire with a multidimensional structure, has been used to evaluate the six psychological well-being dimensions conceptualized by Carol Ryff (autonomy, environmental mastery, personal growth, positive relationships, purpose in life, self-acceptance), which include 14 items each. Every item is defined in terms of high or low agreement on a 6-point Likert scale (ranging from 1 to 6); therefore each scale score may range from 14 to 84, with higher scores corresponding to greater psychological well-being.
  scores on a scale
    Autonomy | 62.20 (9.18) | 61.80 (9.25) | 62 (9.17)
    Environmental mastery | 55.28 (11.52) | 55.32 (10.65) | 55.30 (11.04)
    Personal growth | 60.48 (9.88) | 56.18 (10.50) | 58.33 (10.37)
    Positive relations with others | 61.26 (13.26) | 60.2 (10.68) | 60.73 (11.99)
    Purpose in life | 56.8 (11.51) | 56.22 (11.59) | 56.51 (11.5)
    Self-acceptance | 54.48 (11.63) | 55.8 (13.68) | 55.14 (12.65)
Depression (DSM) [Count of Participants; unit: Participants] — The presence of clinical depression (Major/minor depression or dysthymia) was assessed by means of the Structured Clinical Interview for DSM-IV-TR Axis I Disorders.(SCID-I), a semistuctured interview designed to be administered by a clinician or trained mental health professional in order to formulate psychiatric diagnoses based on the Diagnostic and Statistical Manual of Mental Disorders (DSM).
  Participants | 35 | 27 | 62
Demoralization (DCPR) [Count of Participants; unit: Participants] — Demoralization was assessed by means of the Semi-Structured Interview based on the Diagnostic Criteria for Psychosomatic Research (DCPR), which is an observer-rated measure including skip questions if the main criteria are not satisfied.
  Participants | 47 | 44 | 91
Clinical Interview for Depression (CID) [Mean (Standard Deviation); unit: scores on a scale] — Paykel's 20-item change version of the Clinical Interview for Depression (CID) allows a comprehensive assessment of affective symptomatology and contains 20 items rated on 7-point scales with specification of each anchor point based on severity, frequency and/or quality of symptoms. It adds a dimensional description of mental suffering to traditional psychiatric nosography (DSM). The total score is obtained by adding each of 20 items and it may range from 20 to 140. The higher the score, the worse the psychological condition.
  scores on a scale | 38.18 (8.48) | 36.2 (8.57) | 37.19 (8.54)

OUTCOME MEASURES:

1. Primary Outcome: Depression and Well-being Improvements After Cognitive-Behavioral Therapy and Well-Being Therapy as Assessed by Changes in Clinical Interview for Depression, Compared to Clinical Management
Description: Paykel's 20-item change version of the Clinical Interview for Depression (CID) allows a comprehensive assessment of affective symptomatology and contains 20 items rated on 7-point scales with specification of each anchor point based on severity, frequency and/or quality of symptoms. It adds a dimensional description of mental suffering to traditional psychiatric nosography (DSM). The total score is obtained by adding each of 20 items and it may range from 20 to 140. The higher the score, the worse the psychological condition.
Time Frame: Pre-Treatment, Immediately Post-Treatment, 3-, 6-, 12-, 30-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- CBT/WBT: Patients treated with Cognitive-Behavioral Therapy in combination with Well-Being Therapy and lifestyle modification (experimental group)
  CBT involves several essential features: identifying and correcting inaccurate thoughts associated with depressed feelings (cognitive restructuring); helping patients to engage more often in enjoyable activities (behavioral activation); enhancing problem-solving skills; providing instruction and guidance in specific strategies for solving problems. The techniques included in WBT may be used in overcoming impairments in environmental mastery, purpose in life, personal growth, autonomy, self-acceptance and positive relations with others.
Arm/Group | CBT/WBT | Clinical Management
Number analyzed (Participants) | 50 | 50
score on a scale
  Pre-treatment | 38.18 (8.48) | 36.20 (8.57)
  Post-treatment | 29.39 (6.55) | 32.30 (7.26)
  3-month follow-up | 30.48 (5.81) | 31.89 (7.11)
  6-month follow-up | 29.89 (5.88) | 30.59 (7.28)
  12-month follow-up | 29.70 (6.51) | 30.03 (7.05)
  30-month follow-up | 30.64 (7.02) | 30.30 (6.82)
Statistical Analysis 1: Comparison: CBT/WBT vs Clinical Management; Test type: Superiority; p = 0.030, Repeated Measures ANOVA; All analyses were performed by using intention-to-treat (ITT) analysis, where missing values were managed by means of multiple imputations procedure

2. Primary Outcome: Depression and Well-being Improvements After Cognitive-Behavioral Therapy and Well-Being Therapy as Assessed by Changes in Symptom Questionnaire ("Anxiety" Subscale), Compared to Clinical Management
Description: Anxious symptoms subscale of Kellner's Symptom Questionnaire (SQ). SQ is a 92-item self-report questionnaire, which yields 4 main scales including 23 items each: "depression", "anxiety", "hostility-irritability" and "somatization". This instrument helps the identification of self-perceived subclinical psychological distress. Answers are dichotomous (YES/NO or TRUE/FALSE) and rated with 0 or 1, therefore each scale score may range from 0 to 23. The higher the total score, the higher the psychological distress.
Time Frame: Pre-Treatment, Immediately Post-Treatment, 3-, 6-, 12-, 30-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT/WBT | Clinical Management
Number analyzed (Participants) | 50 | 50
score on a scale
  ANXIETY (SQ) Pre-treatment | 8.60 (4.73) | 7.24 (4.67)
  ANXIETY (SQ) Post-treatment | 7.04 (5.23) | 6.39 (4.41)
  ANXIETY (SQ) 3-month follow-up | 6.60 (4.87) | 6.13 (4.21)
  ANXIETY (SQ) 6-month follow-up | 6.67 (4.19) | 7.10 (5.14)
  ANXIETY (SQ) 12-month follow-up | 6.62 (4.51) | 6.33 (5.09)
  ANXIETY (SQ) 30-month follow-up | 6.00 (4.35) | 5.69 (4.07)
Statistical Analysis 1: Comparison: CBT/WBT vs Clinical Management; Test type: Superiority; p > 0.05, Repeated Measures ANOVA; [statistical method as in outcome 1, analysis 1]

3. Primary Outcome: Depression and Well-being Improvements After Cognitive-behavioral Therapy and Well-Being Therapy Assessed by Changes in Psychological Well-Being Scales ("Autonomy" Dimension), Compared to Clinical Management
Description: Autonomy dimension of the Psychological Well-Being scales (PWB). PWB, an 84-item questionnaire with a multidimensional structure, has been used to evaluate the six psychological well-being dimensions conceptualized by Carol Ryff (autonomy, environmental mastery, personal growth, positive relationships, purpose in life, self-acceptance), which include 14 items each. Every item is defined in terms of high or low agreement on a 6-point Likert scale (ranging from 1 to 6); therefore each scale score may range from 14 to 84, with higher scores corresponding to greater psychological well-being.
Time Frame: Pre-Treatment, Immediately Post-Treatment, 3-, 6-, 12-, 30-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT/WBT | Clinical Management
Number analyzed (Participants) | 50 | 50
score on a scale
  AUTONOMY (PWB) Pre-treatment | 62.20 (9.18) | 61.80 (9.25)
  AUTONOMY (PWB) Post-treatment | 64.58 (9.42) | 62.82 (8.77)
  AUTONOMY (PWB) 3-month follow-up | 64.54 (9.24) | 63.20 (8.51)
  AUTONOMY (PWB) 6-month follow-up | 64.40 (9.12) | 63.21 (9.00)
  AUTONOMY (PWB) 12-month follow-up | 65.50 (8.53) | 64.57 (9.34)
  AUTONOMY (PWB) 30-month follow-up | 64.93 (9.67) | 63.71 (9.26)
Statistical Analysis 1: Comparison: CBT/WBT vs Clinical Management; Test type: Superiority; p > 0.05, Repeated Measures ANOVA; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Number of Participants With Hospitalizations for Cardiac Problems, Revascularization, Recurrent Nonfatal Myocardial Infarction or Cardiac Mortality at 30-month Follow-up.
Description: Frequencies of negative cardiac outcomes, such as re-hospitalizations due to cardiac complications, acute myocardial infarction, unstable angina, angioplasty, cardiac surgery, and cardiac mortality occuring after the first episode of ACS.
Time Frame: 30-month follow-up post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | CBT/WBT | Clinical Management
Number analyzed (Participants) | 50 | 50
Participants
  Non-fatal cardiac events | 8 | 5
  Cardiac death | 1 | 1
  No events | 41 | 44
Statistical Analysis 1: Comparison: CBT/WBT vs Clinical Management; Test type: Superiority; p > 0.05, Kaplan-Meier Survival analysis

5. Primary Outcome: Depression and Well-being Improvements After Cognitive-Behavioral Therapy and Well-Being Therapy as Assessed by Changes in Symptom Questionnaire ("Depression" Subscale), Compared to Clinical Management
Description: Depressive symptoms subscale of Kellner's Symptom Questionnaire (SQ). SQ is a 92-item self-report questionnaire, which yields 4 main scales including 23 items each: "depression", "anxiety", "hostility-irritability" and "somatization". This instrument helps the identification of self-perceived subclinical psychological distress. Answers are dichotomous (YES/NO or TRUE/FALSE) and rated with 0 or 1, therefore each scale score may range from 0 to 23. The higher the total score, the higher the psychological distress.
Time Frame: Pre-Treatment, Immediately Post-Treatment, 3-, 6-, 12-, 30-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT/WBT | Clinical Management
Number analyzed (Participants) | 50 | 50
score on a scale
  DEPRESSION (SQ) Pre-treatment | 7.92 (4.77) | 6.90 (4.87)
  DEPRESSION (SQ) Post-treatment | 7.21 (5.42) | 5.94 (4.22)
  DEPRESSION (SQ) 3-month follow-up | 6.38 (5.03) | 5.83 (4.75)
  DEPRESSION (SQ) 6-month follow-up | 7.06 (5.22) | 6.80 (5.45)
  DEPRESSION (SQ) 12-month follow-up | 6.91 (5.08) | 6.22 (5.09)
  DEPRESSION (SQ) 30-month follow-up | 5.99 (4.64) | 5.83 (4.18)
Statistical Analysis 1: Comparison: CBT/WBT vs Clinical Management; Test type: Superiority; p > 0.05, Repeated Measures ANOVA; [statistical method as in outcome 1, analysis 1]

6. Primary Outcome: Depression and Well-being Improvements After Cognitive-Behavioral Therapy and Well-Being Therapy as Assessed by Changes in Symptom Questionnaire ("Somatization" Subscale), Compared to Clinical Management
Description: Somatic symptoms subscale of Kellner's Symptom Questionnaire (SQ). SQ is a 92-item self-report questionnaire, which yields 4 main scales including 23 items each: "depression", "anxiety", "hostility-irritability" and "somatization". This instrument helps the identification of self-perceived subclinical psychological distress. Answers are dichotomous (YES/NO or TRUE/FALSE) and rated with 0 or 1, therefore each scale score may range from 0 to 23. The higher the total score, the higher the psychological distress.
Time Frame: Pre-Treatment, Immediately Post-Treatment, 3-, 6-, 12-, 30-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT/WBT | Clinical Management
Number analyzed (Participants) | 50 | 50
score on a scale
  SOMATIZATION (SQ) Pre-treatment | 9.82 (5.65) | 7.82 (5.12)
  SOMATIZATION (SQ) Post-treatment | 8.80 (5.73) | 8.24 (4.90)
  SOMATIZATION (SQ) 3-month follow-up | 8.67 (5.42) | 7.87 (4.58)
  SOMATIZATION (SQ) 6-month follow-up | 8.96 (5.02) | 8.15 (5.64)
  SOMATIZATION (SQ) 12-month follow-up | 9.49 (5.19) | 7.90 (5.38)
  SOMATIZATION (SQ) 30-month follow-up | 8.17 (5.00) | 7.61 (4.72)
Statistical Analysis 1: Comparison: CBT/WBT vs Clinical Management; Test type: Superiority; p > 0.05, Repeated Measures ANOVA; [statistical method as in outcome 1, analysis 1]

7. Primary Outcome: Depression and Well-being Improvements After Cognitive-Behavioral Therapy and Well-Being Therapy as Assessed by Changes in Symptom Questionnaire ("Hostility" Subscale), Compared to Clinical Management
Description: Hostility symptoms subscale of Kellner's Symptom Questionnaire (SQ). SQ is a 92-item self-report questionnaire, which yields 4 main scales including 23 items each: "depression", "anxiety", "hostility-irritability" and "somatization". This instrument helps the identification of self-perceived subclinical psychological distress. Answers are dichotomous (YES/NO or TRUE/FALSE) and rated with 0 or 1, therefore each scale score may range from 0 to 23. The higher the total score, the higher the psychological distress.
Time Frame: Pre-Treatment, Immediately Post-Treatment, 3-, 6-, 12-, 30-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT/WBT | Clinical Management
Number analyzed (Participants) | 50 | 50
score on a scale
  HOSTILITY (SQ) Pre-treatment | 4.70 (4.00) | 5.34 (4.36)
  HOSTILITY (SQ) Post-treatment | 5.19 (4.96) | 4.12 (3.78)
  HOSTILITY (SQ) 3-month follow-up | 5.18 (4.46) | 4.71 (3.92)
  HOSTILITY (SQ) 6-month follow-up | 4.41 (3.71) | 6.01 (4.73)
  HOSTILITY (SQ) 12-month follow-up | 5.32 (4.71) | 5.17 (4.14)
  HOSTILITY (SQ) 30-month follow-up | 3.81 (3.37) | 4.56 (4.11)
Statistical Analysis 1: Comparison: CBT/WBT vs Clinical Management; Test type: Superiority; p = 0.013, Repeated Measures ANOVA; [statistical method as in outcome 1, analysis 1]

8. Primary Outcome: Depression and Well-being Improvements After Cognitive-behavioral Therapy and Well-Being Therapy Assessed by Changes in Psychological Well-Being Scales ("Environmental Mastery" Dimension), Compared to Clinical Management
Description: Environmental mastery dimension of the Psychological Well-Being scales (PWB). PWB, an 84-item questionnaire with a multidimensional structure, has been used to evaluate the six psychological well-being dimensions conceptualized by Carol Ryff (autonomy, environmental mastery, personal growth, positive relationships, purpose in life, self-acceptance), which include 14 items each. Every item is defined in terms of high or low agreement on a 6-point Likert scale (ranging from 1 to 6); therefore each scale score may range from 14 to 84, with higher scores corresponding to greater psychological well-being.
Time Frame: Pre-Treatment, Immediately Post-Treatment, 3-, 6-, 12-, 30-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT/WBT | Clinical Management
Number analyzed (Participants) | 50 | 50
score on a scale
  ENVIRONMENTAL MASTERY (PWB) Pre-treatment | 55.28 (11.52) | 55.32 (10.65)
  ENVIRONMENTAL MASTERY (PWB) Post-treatment | 57.33 (12.93) | 56.69 (8.81)
  ENVIRONMENTAL MASTERY (PWB) 3-month follow-up | 59.48 (11.32) | 57.81 (10.15)
  ENVIRONMENTAL MASTERY (PWB) 6-month follow-up | 58.02 (11.83) | 57.51 (8.78)
  ENVIRONMENTAL MASTERY (PWB) 12-month follow-up | 58.36 (12.15) | 58.03 (11.19)
  ENVIRONMENTAL MASTERY (PWB) 30-month follow-up | 58.69 (10.97) | 58.81 (8.10)
Statistical Analysis 1: Comparison: CBT/WBT vs Clinical Management; Test type: Superiority; p > 0.05, Repeated Measures ANOVA; [statistical method as in outcome 1, analysis 1]

9. Primary Outcome: Depression and Well-being Improvements After Cognitive-behavioral Therapy and Well-Being Therapy Assessed by Changes in Psychological Well-Being Scales ("Personal Growth" Dimension), Compared to Clinical Management
Description: Personal growth dimension of the Psychological Well-Being scales (PWB). PWB, an 84-item questionnaire with a multidimensional structure, has been used to evaluate the six psychological well-being dimensions conceptualized by Carol Ryff (autonomy, environmental mastery, personal growth, positive relationships, purpose in life, self-acceptance), which include 14 items each. Every item is defined in terms of high or low agreement on a 6-point Likert scale (ranging from 1 to 6); therefore each scale score may range from 14 to 84, with higher scores corresponding to greater psychological well-being.
Time Frame: Pre-Treatment, Immediately Post-Treatment, 3-, 6-, 12-, 30-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT/WBT | Clinical Management
Number analyzed (Participants) | 50 | 50
score on a scale
  PERSONAL GROWTH (PWB) Pre-treatment | 60.48 (9.88) | 56.18 (10.50)
  PERSONAL GROWTH (PWB) Post-treatment | 61.46 (9.92) | 56.54 (8.70)
  PERSONAL GROWTH (PWB) 3-month follow-up | 61.95 (9.91) | 56.67 (9.65)
  PERSONAL GROWTH (PWB) 6-month follow-up | 60.79 (9.58) | 57.10 (8.90)
  PERSONAL GROWTH (PWB) 12-month follow-up | 60.55 (9.54) | 57.64 (10.24)
  PERSONAL GROWTH (PWB) 30-month follow-up | 59.94 (9.34) | 57.00 (8.85)
Statistical Analysis 1: Comparison: CBT/WBT vs Clinical Management; Test type: Superiority; p > 0.05, Repeated Measures ANOVA; [statistical method as in outcome 1, analysis 1]

10. Primary Outcome: Depression and Well-being Improvements After Cognitive-behavioral Therapy and Well-Being Therapy Assessed by Changes in Psychological Well-Being Scales ("Positive Relations" Dimension), Compared to Clinical Management
Description: Positive relations dimension of the Psychological Well-Being scales (PWB). PWB, an 84-item questionnaire with a multidimensional structure, has been used to evaluate the six psychological well-being dimensions conceptualized by Carol Ryff (autonomy, environmental mastery, personal growth, positive relationships, purpose in life, self-acceptance), which include 14 items each. Every item is defined in terms of high or low agreement on a 6-point Likert scale (ranging from 1 to 6); therefore each scale score may range from 14 to 84, with higher scores corresponding to greater psychological well-being.
Time Frame: Pre-Treatment, Immediately Post-Treatment, 3-, 6-, 12-, 30-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT/WBT | Clinical Management
Number analyzed (Participants) | 50 | 50
score on a scale
  POSITIVE RELATIONS (PWB) Pre-treatment | 61.26 (13.26) | 60.20 (10.68)
  POSITIVE RELATIONS (PWB) Post-treatment | 61.82 (13.50) | 59.90 (10.93)
  POSITIVE RELATIONS (PWB) 3-month follow-up | 61.88 (12.86) | 59.93 (12.13)
  POSITIVE RELATIONS (PWB) 6-month follow-up | 60.60 (13.08) | 58.78 (10.82)
  POSITIVE RELATIONS (PWB) 12-month follow-up | 61.27 (12.08) | 58.95 (11.54)
  POSITIVE RELATIONS (PWB) 30-month follow-up | 60.48 (11.60) | 60.56 (10.78)
Statistical Analysis 1: Comparison: CBT/WBT vs Clinical Management; Test type: Superiority; p > 0.05, Repeated Measures ANOVA; [statistical method as in outcome 1, analysis 1]

11. Primary Outcome: Depression and Well-being Improvements After Cognitive-behavioral Therapy and Well-Being Therapy Assessed by Changes in Psychological Well-Being Scales ("Purpose in Life" Dimension), Compared to Clinical Management
Description: Purpose in life dimension of the Psychological Well-Being scales (PWB). PWB, an 84-item questionnaire with a multidimensional structure, has been used to evaluate the six psychological well-being dimensions conceptualized by Carol Ryff (autonomy, environmental mastery, personal growth, positive relationships, purpose in life, self-acceptance), which include 14 items each. Every item is defined in terms of high or low agreement on a 6-point Likert scale (ranging from 1 to 6); therefore each scale score may range from 14 to 84, with higher scores corresponding to greater psychological well-being.
Time Frame: Pre-Treatment, Immediately Post-Treatment, 3-, 6-, 12-, 30-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT/WBT | Clinical Management
Number analyzed (Participants) | 50 | 50
score on a scale
  PURPOSE IN LIFE (PWB) Pre-treatment | 56.80 (11.51) | 56.22 (11.59)
  PURPOSE IN LIFE (PWB) Post-treatment | 57.31 (11.21) | 54.97 (9.41)
  PURPOSE IN LIFE (PWB) 3-month follow-up | 58.35 (10.09) | 55.47 (10.32)
  PURPOSE IN LIFE (PWB) 6-month follow-up | 57.88 (10.85) | 55.96 (10.12)
  PURPOSE IN LIFE (PWB) 12-month follow-up | 57.42 (9.81) | 55.63 (10.82)
  PURPOSE IN LIFE (PWB) 30-month follow-up | 57.63 (9.70) | 57.76 (8.16)
Statistical Analysis 1: Comparison: CBT/WBT vs Clinical Management; Test type: Superiority; p > 0.05, Repeated Measures ANOVA; [statistical method as in outcome 1, analysis 1]

12. Primary Outcome: Depression and Well-being Improvements After Cognitive-behavioral Therapy and Well-Being Therapy Assessed by Changes in Psychological Well-Being Scales ("Self-acceptance" Dimension), Compared to Clinical Management
Description: Self-acceptance dimension of the Psychological Well-Being scales (PWB). PWB, an 84-item questionnaire with a multidimensional structure, has been used to evaluate the six psychological well-being dimensions conceptualized by Carol Ryff (autonomy, environmental mastery, personal growth, positive relationships, purpose in life, self-acceptance), which include 14 items each. Every item is defined in terms of high or low agreement on a 6-point Likert scale (ranging from 1 to 6); therefore each scale score may range from 14 to 84, with higher scores corresponding to greater psychological well-being.
Time Frame: Pre-Treatment, Immediately Post-Treatment, 3-, 6-, 12-, 30-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT/WBT | Clinical Management
Number analyzed (Participants) | 50 | 50
score on a scale
  SELF-ACCEPTANCE (PWB) Pre-treatment | 54.58 (11.63) | 55.80 (13.68)
  SELF-ACCEPTANCE (PWB) Post-treatment | 55.70 (14.36) | 56.03 (11.52)
  SELF-ACCEPTANCE (PWB) 3-month follow-up | 57.59 (13.51) | 57.86 (12.84)
  SELF-ACCEPTANCE (PWB) 6-month follow-up | 55.83 (14.19) | 58.32 (12.39)
  SELF-ACCEPTANCE (PWB) 12-month follow-up | 56.66 (11.92) | 59.69 (13.38)
  SELF-ACCEPTANCE (PWB) 30-month follow-up | 56.15 (13.90) | 59.94 (10.52)
Statistical Analysis 1: Comparison: CBT/WBT vs Clinical Management; Test type: Superiority; p > 0.05, Repeated Measures ANOVA; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From pre-treatment (baseline) to 30-month follow-up after the end of the interventions (both CBT/WBT and CM)
Description: Re-hospitalizations due to cardiac complications, acute myocardial infarction, unstable angina, angioplasty and cardiac surgery occured after the first episode of ACS
Arm/Group | CBT/WBT | Clinical Management
All-Cause Mortality (participants affected / at risk) | 1/50 | 1/50
Serious Adverse Events (participants affected / at risk) | 9/50 | 6/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CBT/WBT (N=50) | Clinical Management (N=50)
Non-fatal cardiac events (Cardiac disorders) | 8 | 5 — Re-hospitalizations due to cardiac complications, acute myocardial infarction, unstable angina, angioplasty and cardiac surgery after the first episode of ACS
Cardiac death (Cardiac disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2009-10-19): https://cdn.clinicaltrials.gov/large-docs/00/NCT00998400/Prot_SAP_000.pdf